CLINICAL TRIAL: NCT02035683
Title: Study of the Role of Metabolic Response Measured by PET/CT Scan After 1 Cycle of Chemotherapy in Patients With Advanced Non Small Cell Lung Cancer (NSCLC)
Brief Title: PET/CT Scan as a Tool to Rationalize the Treatment of of Advanced NSCLC Patients Undergoing First Chemotherapy
Acronym: PETRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PETRA
Record Dates: First submitted 2014-01-07; First posted 2014-01-14 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Non-small Cell Lung Cancer Stage IIIB
Keywords: metabolic response; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Advanced NSCLC patients undergoing first-line chemotherapy (Other): single cohort
  Interventions: Procedure: PET/CT

INTERVENTIONS:
Procedure: PET/CT — PET/CT scan at baseline and 3 weeks after first cycle chemotherapy

SUMMARY:
The purpose of this study is to test whether an early metabolic response, measured by PET/CT scan after the first cycle of chemotherapy, is able to predict which patients with advanced NSCLC have a better prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cytologically or histologically confirmed non-small cell lung cancer.
* Metastatic (stage IV, both M1A or M1B) or locally advanced (stage IIIB, with metastasis to supraclavicular nodes) according to TNM VII edition.
* Both patients at first diagnosis or those with disease recurrence after initial surgery are eligible.
* At least one target or non-target lesion according to RECIST revised version 1.1.
* Age > or = 18 years .
* ECOG PS 0-2.
* Life expectancy > 3 months.
* Signed informed consent.

Exclusion Criteria:

* Uncontrolled diabetes (glucose > 200 mg/dl
* EGFR mutation, for those patients who have had testing done. (EGFR test is not required for participation in the study, but may be conducted as part of normal clinical practice, and patients with EGFR mutation would not be candidate for first-line chemotherapy.)
* Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer or surgically resected prostate cancer with normal PSA).
* Pregnant or lactating females.
* Previous medical therapy for metastatic disease (prior surgery, radiation therapy are permitted, as well as adjuvant medical therapy completed at least 6 months prior to study entry).
* Any poorly controlled illness (including active infections, significant hepatic, renal, metabolic or cardiac disease, myocardial infarction within previous 12 months) that may, according to physician's judgement, interfere with the patient's ability to undergo chemotherapy and/or the examinations within the study protocol
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-10; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline in highest value SUVmax (maximum standardized uptake values in PET/CT scan) | one year
  To validate as prognostic factor, in terms of overall survival,early metabolic response, defined as a reduction of more than 50% of the highest value of SUVmax recorded at PET/CT scan after one cycle of chemotherapy, compared to the highest value of SUVmax recorded baseline examination

SECONDARY OUTCOMES:
Change from baseline in SUVmaxsum, TLGmax and TLGmaxsum | one year
  to describe and validate early metabolic response as a prognostic factor (in terms of overall survival), using the sum of the SUVmax (SUVmaxsum) , the highest value of TLG (TLGmax), the sum of TLG ( TLGmaxsum).
correlation among SUVmax, SUVmaxsum, TLGmax, TLGsum with progression-free survival | one year
  prognostic role of early metabolic response (defined according the above reported 4 parameters) in terms of progression free survival after a first line chemotherapy
correlation among SUVmax, SUVmaxsum, TLGmax, TLGsum with objective response | 3 months
  To describe the association between early metabolic response (defined according the above reported 4 parameters) and objective response according RECIST criteria, measured after 3 cycles of chemotherapy
overall survival | one year
progression free survival | 12 months
objective response | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Secondo Lastoria, M.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute Naples, Italy; Director Clinical Trials Unit; Ciro Gallo, M.D., Ph.D, Principal Investigator — Second University of Naples, Italy; Chair of Medical Statistics; Massimo Di Maio, M.D., Principal Investigator — National Cancer Institute, Naples; Alessandro Morabito, M.D., Principal Investigator — National Cancer Institute, Naples; Gaetano Rocco, M.D., Principal Investigator — National Cancer Institute, Naples
Locations (1):
- Istituto Nazionale dei Tumori, Napoli, Italy